CLINICAL TRIAL: NCT02699827
Title: Adding Magnesium Sulphate to Epidural Levobupivacaine in Elective Caesarian Section for Patients With Preeclampsia
Brief Title: Adding MgSO4 to Epidural Levobupivacaine in CS for Patients With Preeclampsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TM1
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Preeclampsia
Keywords: Levobupivacaine; Magnesium; Preeclampsia; Epidural
MeSH Terms: conditions — Pre-Eclampsia | interventions — Levobupivacaine; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium sulphate group (Active Comparator): Patients will receive epidural levobupivacaine hydrochloride + magnesium sulphate
  Interventions: Drug: Levobupivacaine hydrochloride; Drug: Magnesium sulphate
- Placebo group (Placebo Comparator): Patients will receive epidural levobupivacaine hydrochloride + saline 0.9%
  Interventions: Drug: Levobupivacaine hydrochloride; Drug: Saline 0.9%

INTERVENTIONS:
Drug: Levobupivacaine hydrochloride — Patients will receive epidural 20 ml levobupivacaine hydrochloride 0.5%
  Other Names: Chirocaine
Drug: Magnesium sulphate — Patients will receive epidural 5 ml magnesium sulphate 10%
  Arms: Magnesium sulphate group
Drug: Saline 0.9% — Patients will receive epidural 5 ml saline 0.9%
  Arms: Placebo group

SUMMARY:
This study aims at evaluating the effect of adding magnesium sulphate epidurally as an adjunct to levobupivacaine on the quality of anesthesia and perioperative pain relief in patients with preeclampsia undergoing elective caesarian section (CS).

DETAILED DESCRIPTION:
Pregnant women with preeclampsia undergoing elective CS in will be included in the study. All patients participating in the study will be randomly divided into two groups; magnesium sulphate group (study group) and placebo group (control group). Patients in the study group will receive epidural 20 ml levobupivacaine hydrochloride 0.5% plus 5 ml magnesium sulphate 10% (500 mg) while patients in the control group will received epidural 20 ml levobupivacaine hydrochloride 0.5% plus 5 ml saline 0.9%.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with preeclampsia undergoing elective CS.

Exclusion Criteria:

* Age < 20 or > 35 years.
* Height < 150 or > 180 cm.
* Body mass index (BMI) > 35 kg/m2.
* Active labor.
* Multifetal pregnancy.
* Fetal distress.
* Medical conditions complicating pregnancy.
* HELLP syndrome.
* Thrombocytopenia.
* Hepatic or renal impairment.
* Pulmonary edema or cyanosis.
* Placenta previa.
* Vaginal bleeding or placental abruption.
* Contraindication for central neuraxial block.
* History of adverse reaction to any study medication.
* History of analgesic use.
* Magnesium therapy.
* Chronic pain syndrome.
* Presence of communication difficulties preventing reliable assessment.
* Refusal to undergo regional anesthesia.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pain-free period | 24 hours after the epidural anesthesia
  The time from reaching sensory block to onset of pain

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Elmetwally, Dr, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University; Reem A Elsharkawy, Dr, Study Director — Mansoura University; Waleed El-refaie, Dr, Study Director — Mansoura University; Alaa Wageeh, Dr, Study Director — Mansoura University; Salwa S Hays, Prof, Study Chair — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided